CLINICAL TRIAL: NCT00248950
Title: A Pilot Study: Changing Multiple Behaviors in Post-Angioplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Mary E. Charlson, MD, Weill Cornell Medical College
Allocation: Non-Randomized | Model: Single Group | Masking: Double
Other Study IDs: N01-HC-25196 (0103-660); N01HC25196 (NIH)
Record Dates: First submitted 2005-11-03; First posted 2005-11-04 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Angioplasty Patients
Keywords: Angioplasty; Behavior Change

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Positive affect induction and /or self affirmation induction

SUMMARY:
We are interested in achieving an empirical test of the two intervention approaches under study. Specifically, we seek to determine the potential differential impact of positive affect induction and self affirmation following the qualitative study phase.

DETAILED DESCRIPTION:
We seek to determine the potential differential impact of positive affect induction and self affirmation following the qualitative study phase.

1. Positive affect induction: We will tests two types of positive affect induction. 1) sending patients a small gift, and 2) reminding patients of positive thoughts about themselves. Gift: Prior to a telephone call, patients in the positive affect condition will receive a small gift. The selection of gifts will be guided, in part, by data obtained from the qualitative study phase. Positive thoughts about themselves: Patients will be asked to describe a time when someone was helpful to them, and they felt good about it , and were nice to them in return.
2. Self affirmation: consists of a series of items reminding people of their core values.
3. Control: Control patients will have neither self affirmation nor gifts. After enrollment, patients will be randomized into four groups: control, the self affirmation, the positive affect gift group and the positive affect positive thought group. Thus, for the positive affect, we will test two different types of positive affect induction.

Follow-up: At two weeks after enrollment all patients will be called to ascertain impact of the pilot intervention.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing coronary artery catheterization who are found to have at least single vessel stenosis and who have had revascularization with angioplasty or coronary artery stenting will be eligible for enrollment. Patients must be able to provide informed consent within the one week after the procedure.

Exclusion Criteria:

1. Patients who are unable to walk several blocks regardless of the reason will be excluded from all the trials (e.g., arthritis, stroke, claudication).
2. Enrollment in other trials designed to modify post-procedure behaviors.
3. Patients who refuse to participate will be excluded.
4. If at any time prior to enrollment in the study, the patient's cardiologist determines that the patient should not participate in this study, the patient will not be enrolled in the trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2004-02; Study Completion 2004-06

PRIMARY OUTCOMES:
Within patient change on the Positive and Negative Affect Scale

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Charlson, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- The New York Presbyterian Hospital-Weill Medical Center, New York, New York, United States